CLINICAL TRIAL: NCT06451705
Title: Comparison Between Pectoral Nerve Block II and Local Anesthesia Infiltration of Isobaric Bupivacaine 0.25% 50 MG on Neutrophil-Lymphocyte Ratio, Interleukin-6 Levels, Pain Intensity, and Post-surgical Opioid Requirements in Modified Radical Mastectomy Patients
Brief Title: Pecs Block vs Local Infiltration in Mastectomy
Acronym: PBLIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasanuddin University (Other)
Responsible Party: Principal Investigator, Jokevin Prasetyadhi, Principal Investigator, Hasanuddin University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 173/UN4.6.4.5.31/PP36/2AZ4
Record Dates: First submitted 2024-05-23; First posted 2024-06-11 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Pain, Postoperative
Keywords: postoperative pain; modified radical mastectomy; peripheral nerve block; local infiltration anesthesia; pectoralis nerve block
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: single-blind randomized trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PECS (Active Comparator): PECS II block before surgery using isobaric bupivacaine 0.25% 20 mL (50 mg)
  Interventions: Drug: PECS II block
- LIA (Active Comparator): Local infiltration anesthesia after completion of surgery using isobaric bupivacaine 0.25% 20 mL (50 mg)
  Interventions: Drug: LIA

INTERVENTIONS:
Drug: PECS II block — Treatment group that received the PECS II block using isobaric bupivacaine 0.5% 50 mg
  Arms: PECS
Drug: LIA — Treatment group that received the local infiltration anesthesia using isobaric bupivacaine 0.5% 50 mg
  Arms: LIA

SUMMARY:
Studied the comparison between PECS II block and LIA on pain intensity, opioid requirements, RNL, and postoperative IL-6 levels in MRM patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-60 years old.
2. Body weight (BW): 50-70 kg.
3. Height (TB): 150-170 cm.
4. Body mass index (BMI): 18.5-29.9 kg/m2.
5. American Society of Anesthesiologists physical status (ASA PS) class I-II.
6. Patients undergoing elective MRM surgery under general anesthesia.

Exclusion Criteria:

1. Patients with contraindications to PECS II block.
2. Patients with contraindications to LIA.
3. Patients with coagulation disorders or receiving anticoagulant therapy.
4. Patients with a history of chronic pain.
5. Patients with a history of allergy to study materials.
6. Patients with a history of previous breast surgery.
7. Patient refuses to participate in the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Concentration of Plasma Interleukin-6 | 1 hour before surgery, 2 hour after surgery, 12 hour after surgery
  in pg/dL
Neutrophil-lymphocyte ratio | 1 hour before surgery, 2 hour after surgery, 12 hour after surgery
  Neutrophil divided by lymphocyte
Pain intensity (Using Numeric Rating Scale) | hour 0, 2, 4, 6, 12, 24
  Scale from 0-10, lower score = better outcome
Rescue opioid requirement | Within 24 hours after surgery
  Using fentanyl at a dose of 0.5-1 μg/kg/IV titrated as needed, in mcg (given if the patient had NRS of >4/10)

SECONDARY OUTCOMES:
Demographic baseline data | baseline (before the surgery)
  Medical record number, age, body weight (in kilogram), height (in centimeter), BMI (in kg/m2), ASA PS class, duration of surgery (in minutes)
Time until first rescue opioid requirement | Within 24 hours after surgery
  in minutes
Nausea and vomiting | Within 24 hours after surgery
  Nausea and vomiting were assessed using a numerical scale (0 = no nausea, 1 = mild nausea, 2 = severe nausea or vomiting once, and 3 = vomiting more than once). If the score was > 2, rescue antiemetics with ondansetron 0.1 mg/IV were given.

CONTACTS AND LOCATIONS:
Locations (1):
- RSUP dr. Wahidin Sudirohusodo, Makassar, South Sulawesi, Indonesia

IPD SHARING:
Plan to Share IPD: No